CLINICAL TRIAL: NCT01876524
Title: Transcranial Random Noise Stimulation in Anterior Cingulate Cortex Reduces Craving Over Dual Pathology Patients
Brief Title: tRNS in Anterior Cingulate Cortex Reduces Craving Over Dual Pathology Patients
Acronym: tRND&SUDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tRNS01072013
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder; Attention Deficit Disorder With Hyperactivity; Bipolar Disorder; Schizophrenia; Personality Disorder
Keywords: Substance Use Disorder; Attention Deficit Disorder With Hyperactivity; Schizophrenia; Bipolar disorder; Personality disorder
MeSH Terms: conditions — Substance-Related Disorders; Attention Deficit Disorder with Hyperactivity; Bipolar Disorder; Schizophrenia; Personality Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tRNS over Anterior Cingulate (Experimental): Dual Pathology (Substance Use Disorder plus another psychiatric trait) 75 patients with diagnosed SUDs plus another psychiatric disorder will be receive tRNS in the disease-specific Anterior Cingulate Cortex (ACC), be studied blindly to evaluate the craving reduction after 35 tRNS sessions.
  Interventions: Device: Transcranial Random Noise Stimulation
- tRNS applied over DLPFC (Experimental): Dual Pathology (Substance Use Disorder plus another psychiatric trait) 75 patients with diagnosed SUDs plus another psychiatric disorder will be receive tRNS in the dorso-lateral-prefrontal-cortex (DLPFC), be studied blindly to evaluate the craving reduction after 35 tRNS sessions.
  Interventions: Device: Transcranial Random Noise Stimulation
- Sham Group (Sham Comparator): 75 patients will be receive tRNS sham 35 sessions.
  Interventions: Device: Transcranial Random Noise Stimulation

INTERVENTIONS:
Device: Transcranial Random Noise Stimulation — Random Noise Stimulation between 100 and 500 Hz and 400-500 microAmperes are applied over head in particular areas
  Other Names: tRNS, tES

SUMMARY:
The purpose of this study is to study the efficacy and security of noninvasive brain stimulation as a new approach for patients with Substance Use Disorders (SUDs) plus other psychiatric conditions like ADHD, Schizophrenia, Bipolar disorder, etc.

DETAILED DESCRIPTION:
Background: There is an intimate relationship between addictive behaviors and other mental disorders, proven by clinical practice and many epidemiological studies, genetic and neuroscience. This gives risk to the diagnosis of Dual Pathology: an addiction and another mental disorder.

Functional neuroimaging studies have shown that anterior cingulate cortex is associated with substance´s dependence and craving. Transcranial random noise stimulation (tRNS) stimulates parts of the brain and can change it´s activity.

Researchers are interested in reduce cravings for substance dependence on patients with Dual Pathology using tRNS in anterior cingulate cortex.

Aims: To determine whether tRNS in anterior cingulate cortex can reduce craving over Dual Pathology patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old and less than 60 years
* Best-practice diagnosed Dual Pathology
* Diagnosed since at least two years prior to enrollment.
* Abuse more than 2 Substances

ExclusionC riteria:

* Serious visual and hearing loss
* Brain injury following cranial trauma
* Other neurological disorders like Parkinson, ME, headache, etc.
* Birth trauma
* Mental retardation
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
AMEN Questionnarie | Following patients during 3 months after Brain noninvasive estimulation
  100 Items Questionnarie subdivided in 5 subscales: basal ganglia, cingulate cortez, temporal cortex, prefrontal cortex and limbic system
Emotional Visual Event Related Potentials | Following patients during 3 months after Brain noninvasive estimulation
  Emotional Visual Event Related Potentials responses (time courses and topographies) and ICA components related with them, identified by Mitsar 201M EEG Amplifier using EEGLab software [ Time Frame: brainwaves patterns following an array of visual stimuli (human faces) during a 22 min. examination ]

SECONDARY OUTCOMES:
CAGE Adapted to Include Drugs (CAGE-AID) | Following 3 months after tRNS brain stimulation
  The CAGE-AID is a sensitive screen for alcohol and drug problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Slow Environment Foundation, Cartagena, Murcia, Spain

REFERENCES:
- [Background] Manni C, Cipollone G, Pallucchini A, Maremmani AGI, Perugi G, Maremmani I. Remarkable Reduction of Cocaine Use in Dual Disorder (Adult Attention Deficit Hyperactive Disorder/Cocaine Use Disorder) Patients Treated with Medications for ADHD. Int J Environ Res Public Health. 2019 Oct 15;16(20):3911. doi: 10.3390/ijerph16203911. PMID 31618876
- [Background] Allenby C, Falcone M, Bernardo L, Wileyto EP, Rostain A, Ramsay JR, Lerman C, Loughead J. Transcranial direct current brain stimulation decreases impulsivity in ADHD. Brain Stimul. 2018 Sep-Oct;11(5):974-981. doi: 10.1016/j.brs.2018.04.016. Epub 2018 Apr 23. PMID 29885858
- [Background] Cubillo A, Halari R, Smith A, Taylor E, Rubia K. A review of fronto-striatal and fronto-cortical brain abnormalities in children and adults with Attention Deficit Hyperactivity Disorder (ADHD) and new evidence for dysfunction in adults with ADHD during motivation and attention. Cortex. 2012 Feb;48(2):194-215. doi: 10.1016/j.cortex.2011.04.007. Epub 2011 Apr 27. PMID 21575934
- [Background] Fonteneau C, Redoute J, Haesebaert F, Le Bars D, Costes N, Suaud-Chagny MF, Brunelin J. Frontal Transcranial Direct Current Stimulation Induces Dopamine Release in the Ventral Striatum in Human. Cereb Cortex. 2018 Jul 1;28(7):2636-2646. doi: 10.1093/cercor/bhy093. PMID 29688276
- [Result] Westwood SJ, Criaud M, Lam SL, Lukito S, Wallace-Hanlon S, Kowalczyk OS, Kostara A, Mathew J, Agbedjro D, Wexler BE, Cohen Kadosh R, Asherson P, Rubia K. Transcranial direct current stimulation (tDCS) combined with cognitive training in adolescent boys with ADHD: a double-blind, randomised, sham-controlled trial. Psychol Med. 2023 Jan;53(2):497-512. doi: 10.1017/S0033291721001859. Epub 2021 Jul 6. PMID 34225830
- [Result] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- See also: Bigdata4brain LLC — https://www.bigdata4brain.com
- See also: Brainmech Foundation — https://www.brainmech.org